CLINICAL TRIAL: NCT06138795
Title: A Phase I, Randomized, Single-blind, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZD2389 After Single and Multiple Ascending Doses to Healthy Participants.
Brief Title: A Single and Multiple Ascending Dose Study to Investigate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZD2389 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: D7930C00001
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Healthy Participants
Keywords: Liver disease; Single ascending dose; Multiple ascending dose
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Intervention Model Description: Placebo-controlled
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Cohort 1: Part A1 - AZD2389 dose 1/placebo oral administration (Experimental): A total of 6 study participants will receive a single dose of AZD2389 and 2 will receive placebo.
  Interventions: Drug: AZD2389; Drug: Placebo
- Cohort 2: Part A1 - AZD2389 dose 2/placebo oral administration (Experimental): A total of 6 study participants will receive a single dose of AZD2389 and 2 will receive placebo.
  Interventions: Drug: AZD2389; Drug: Placebo
- Cohort 3: Part A1 - AZD2389 dose 3 /placebo oral administration (Experimental): A total of 6 study participants will receive a single dose of AZD2389 and 2 will receive placebo.
  Interventions: Drug: AZD2389; Drug: Placebo
- Cohort 4: Part A1 - AZD2389 dose 4 /placebo oral administration (Experimental): A total of 6 study participants will receive a single dose of AZD2389 and 2 will receive placebo.
  Interventions: Drug: AZD2389; Drug: Placebo
- Cohort 5: Part A1 - AZD2389 dose 5 /placebo oral administration (Experimental): A total of 6 study participants will receive a single dose of AZD2389 and 2 will receive placebo.
  Interventions: Drug: AZD2389; Drug: Placebo
- Cohort 6: Part A1 - AZD2389 dose 6 oral administration (Experimental): A total of 6 study participants will receive a single dose of AZD2389.
  Interventions: Drug: AZD2389
- Cohort 7: Part A2 - AZD2389 dose 7 /placebo oral administration (Experimental): A total of 6 study participants will receive a single dose of AZD2389 and 2 will receive placebo.
  Interventions: Drug: AZD2389; Drug: Placebo
- Cohort 8: Part A2 - AZD2389 dose 8 /placebo oral administration (Experimental): A total of 6 study participants will receive a single dose of AZD2389 and 2 will receive placebo.
  Interventions: Drug: AZD2389; Drug: Placebo
- Cohort 9: Part A2 - AZD2389 dose 9 /placebo oral administration (Experimental): A total of 6 study participants will receive a single dose of AZD2389 and 2 will receive placebo.
  Interventions: Drug: AZD2389; Drug: Placebo
- Cohort 10: Part A3 - AZD2389 dose 10 /placebo oral administration (Experimental): A total of 6 study participants will receive a single dose of AZD2389 and 2 will receive placebo.
  Interventions: Drug: AZD2389; Drug: Placebo
- Cohort 11: Part B1 - AZD2389 dose 11 /placebo oral administration (Experimental): A total of 6 study participants will receive multiple doses of AZD2389 and 2 will receive placebo.
  Interventions: Drug: AZD2389; Drug: Placebo
- Cohort 12: Part B1 - AZD2389 dose 12 /placebo oral administration (Experimental): A total of 6 study participants will receive multiple doses of AZD2389 and 2 will receive placebo.
  Interventions: Drug: AZD2389; Drug: Placebo
- Cohort 13: Part B1 - AZD2389 dose 13 /placebo oral administration (Experimental): A total of 6 study participants will receive multiple doses of AZD2389 and 2 will receive placebo.
  Interventions: Drug: AZD2389; Drug: Placebo
- Cohort 14: Part B2- AZD2389 dose 14/placebo oral administration (Experimental): A total of 6 study participants will receive multiple doses of AZD2389 and 2 will receive placebo.
  Interventions: Drug: AZD2389; Drug: Placebo

INTERVENTIONS:
Drug: AZD2389 — Participants will receive AZD2389 orally as a single ascending dose or multiple ascending dose.
Drug: Placebo — Participants will receive placebo matching the AZD2389 dose orally as a single ascending dose or multiple ascending dose.
  Arms: Cohort 10: Part A3 - AZD2389 dose 10 /placebo oral administration; Cohort 11: Part B1 - AZD2389 dose 11 /placebo oral administration; Cohort 12: Part B1 - AZD2389 dose 12 /placebo oral administration; Cohort 13: Part B1 - AZD2389 dose 13 /placebo oral administration; Cohort 14: Part B2- AZD2389 dose 14/placebo oral administration; Cohort 1: Part A1 - AZD2389 dose 1/placebo oral administration; Cohort 2: Part A1 - AZD2389 dose 2/placebo oral administration; Cohort 3: Part A1 - AZD2389 dose 3 /placebo oral administration; Cohort 4: Part A1 - AZD2389 dose 4 /placebo oral administration; Cohort 5: Part A1 - AZD2389 dose 5 /placebo oral administration; Cohort 7: Part A2 - AZD2389 dose 7 /placebo oral administration; Cohort 8: Part A2 - AZD2389 dose 8 /placebo oral administration; Cohort 9: Part A2 - AZD2389 dose 9 /placebo oral administration

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of AZD2389 following single and multiple dose administration (SAD/MAD) to healthy participants.

DETAILED DESCRIPTION:
This is a Phase I, First In Human (FIH), randomized, single-blind, placebo-controlled, single and multiple ascending dose study in healthy male and/or female participants of non-childbearing potential including healthy participants of Chinese and Japanese ethnicity performed at a single center.

The study consists of 2 parts: Part A and Part B. Part A has been planned to be conducted with 78 participants and Part B has been planned to be conducted with 32 participants.

Each participant in Part A and Part B will be involved in the study for up to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female (of non-childbearing potential) participants with suitable veins for cannulation or repeated venipuncture.
* For the healthy Japanese cohorts (Parts A2 and B2): healthy participants are to be Japanese (e.g., natives of Japan or Japanese Americans), defined as having both parents and 4 grandparents who are Japanese. This includes healthy second and third generation participants of Japanese descent whose parents or grandparents are living in a country other than Japan.
* For the healthy Chinese cohort (Part A3): healthy participants are to be Chinese defined as having both parents and 4 grandparents who are ethnically Chinese. This includes second and third generation Chinese whose parents or grandparents are living in a country other than China.

Exclusion Criteria:

* Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP.
* Known or suspected history of alcohol or drug abuse and smokers.
* Plasma donation within one month of the Screening Visit or any blood donation/blood loss > 500 mL during the 3 months prior to the Screening Visit.
* History of coagulation or bleeding disorders or use of anti-platelets/anti-coagulants during the 3 months prior to the Screening Visit, as judged by the investigator.
* History of hypersensitivity as judged by the investigator, to drugs with a similar chemical structure or class.
* History of severe dermatological disorders, eg, bullous pemphigoid or Stevens-Johnson syndrome, or clinically significant new or healing wounds in areas of the body not always covered by clothing such as face, forearm, and lower leg, as judged by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2025-08-24 (Actual); Study Completion 2025-08-24 (Actual)

PRIMARY OUTCOMES:
Part A (SAD): Number of participants with adverse events (AE) and serious adverse events (SAE) | Day ≤ -28 (Only SAE), Day -1 (Only SAE), Days 1 and 2, Day 8 Post-dose (± 1 day)
  To assess the safety and tolerability of AZD2389 following oral administration of single ascending doses in healthy participants, including Japanese and Chinese participants.
Part B (MAD): Number of participants with AE and SAE | Day ≤ -28 (Only SAE), Day -1 (Only SAE), Days 1 to 12, Day 17 (± 1 day)
  To assess the safety and tolerability of AZD2389 following oral administration of multiple ascending doses in healthy participants, including Japanese participants.

SECONDARY OUTCOMES:
Part A (SAD): Plasma concentrations of AZD2389 | Day 1 and Day 2
  To characterize the plasma concentration of AZD2389 after single oral dosing in healthy participants, including Japanese and Chinese participants.
Part A (SAD): Urine concentrations of AZD2389 | Day 1 and Day 2
  To characterize the urine concentration of AZD2389 after single oral dosing in healthy participants, including Japanese and Chinese participants.
Part A (SAD): Terminal rate constant (λz) | Day 1 and Day 2
  To characterize the λz of AZD2389 after single oral dosing in healthy participants, including Japanese and Chinese participants.
Part A (SAD): Cumulative amount of unchanged drug excreted into urine from time t1 to time t2 [Ae(t1-t2)] | Day 1 and Day 2
  To characterize the Ae(t1-t2) of AZD2389 after single oral dosing in healthy participants, including Japanese and Chinese participants.
Part A (SAD): Area under plasma concentration time curve from zero to infinity (AUCinf) | Day 1 and Day 2
  To characterize the AUCinf of AZD2389 after single oral dosing in healthy participants, including Japanese and Chinese participants.
Part A (SAD): Dose normalized AUCinf (AUCinf/D) | Day 1 and Day 2
  To characterize the AUCinf/D of AZD2389 after single oral dosing in healthy participants, including Japanese and Chinese participants.
Part A (SAD): Area under concentration curve from time 0 to the last quantifiable concentration (AUClast) | Day 1 and Day 2
  To characterize the AUClast of AZD2389 after single oral dosing in healthy participants, including Japanese and Chinese participants.
Part A (SAD): Dose normalized AUClast (AUClast/D) | Day 1 and Day 2
  To characterize the AUClast/D of AZD2389 after single oral dosing in healthy participants, including Japanese and Chinese participants.
Part A (SAD): Apparent total body clearance of drug (CL/F) | Day 1 and Day 2
  To characterize the CL/F of AZD2389 after single oral dosing in healthy participants, including Japanese and Chinese participants.
Part A (SAD): Maximum observed plasma (peak) drug concentration (Cmax) | Day 1 and Day 2
  To characterize the Cmax of AZD2389 after single oral dosing in healthy participants, including Japanese and Chinese participants.
Part A (SAD): Dose normalized Cmax (Cmax/D) | Day 1 and Day 2
  To characterize the Cmax/D of AZD2389 after single oral dosing in healthy participants, including Japanese and Chinese participants.
Part A (SAD): Renal clearance (CLR) | Day 1 and Day 2
  To characterize the CLR of AZD2389 after single oral dosing in healthy participants, including Japanese and Chinese participants.
Part A (SAD): Individual and cumulative percentage of dose excreted unchanged in urine from time t1 to time t2 [fe(t1-t2)] | Day 1 and Day 2
  To characterize the fe(t1-t2) of AZD2389 after single oral dosing in healthy participants, including Japanese and Chinese participants.
Part A (SAD): Mean residence time (MRTinf) | Day 1 and Day 2
  To characterize the MRTinf of AZD2389 after single oral dosing in healthy participants, including Japanese and Chinese participants.
Part A (SAD): Apparent terminal elimination half-life (t½λz) | Day 1 and Day 2
  To characterize the t½λz of AZD2389 after single oral dosing in healthy participants, including Japanese and Chinese participants.
Part A (SAD): Time of last quantifiable concentration (tlast) | Day 1 and Day 2
  To characterize the tlast of AZD2389 after single oral dosing in healthy participants, including Japanese and Chinese participants.
Part A (SAD): Time to reach peak or maximum observed concentration (tmax) | Day 1 and Day 2
  To characterize the tmax of AZD2389 after single oral dosing in healthy participants, including Japanese and Chinese participants.
Part A (SAD): Apparent volume of distribution based on the terminal phase (Vz/F) | Day 1 and Day 2
  To characterize the Vz/F of AZD2389 after single oral dosing in healthy participants, including Japanese and Chinese participants.
Part A (SAD): Change in PD biomarkers over time | Day 1 and Day 2
  To characterize the percentage change in PD biomarkers over time compared to baseline of AZD2389 after single oral dosing in healthy participants, including Japanese and Chinese participants.
Part B (MAD): Plasma concentrations of AZD2389 | Day 1 to Day 12
  To characterize the plasma concentration of AZD2389 following oral administration of multiple ascending doses in healthy participants, including Japanese participants.
Part B (MAD): Urine concentrations of AZD2389 | Day 1 and Days 10 to 12
  To characterize the urine concentration of AZD2389 following oral administration of multiple ascending doses in healthy participants, including Japanese participants.
Part B (MAD): Terminal rate constant (λz) | Day 1 to Day 12
  To characterize the λz of AZD2389 following oral administration of multiple ascending doses in healthy participants, including Japanese participants.
Part B (MAD): Cumulative amount of unchanged drug excreted into urine from time t1 to time t2 [Ae(t1-t2)] | Day 1 and Days 10 to 12
  To characterize the Ae(t1-t2) of AZD2389 following oral administration of multiple ascending doses in healthy participants, including Japanese participants.
Part B (MAD): Area under concentration curve from time 0 to the last quantifiable concentration (AUClast) | Day 1 to Day 12
  To characterize the AUClast of AZD2389 following oral administration of multiple ascending doses in healthy participants, including Japanese participants.
Part B (MAD): Area under the concentration-time curve in the dose interval (AUCtau) | Day 1 to Day 12
  To characterize the AUCtau of AZD2389 following oral administration of multiple ascending doses in healthy participants, including Japanese participants.
Part B (MAD): Dose normalized AUCtau (AUCtau/D) | Day 1 to Day 12
  To characterize the AUCtau/D of AZD2389 following oral administration of multiple ascending doses in healthy participants, including Japanese participants.
Part B (MAD): Dose normalized AUClast (AUClast/D) | Day 1 to Day 12
  To characterize the AUClast/D of AZD2389 following oral administration of multiple ascending doses in healthy participants, including Japanese participants.
Part B (MAD): Apparent total body clearance of drug (CL/F) | Day 1 and Days 10 to 12
  To characterize the CL/F of AZD2389 following oral administration of multiple ascending doses in healthy participants, including Japanese participants.
Part B (MAD): Renal clearance (CLR) | Day 1 and Days 10 to 12
  To characterize the CLR of AZD2389 following oral administration of multiple ascending doses in healthy participants, including Japanese participants.
Part B (MAD): Maximum observed plasma (peak) drug concentration (Cmax) | Day 1 to Day 12
  To characterize the Cmax of AZD2389 following oral administration of multiple ascending doses in healthy participants, including Japanese participants.
Part B (MAD): Dose normalized Cmax (Cmax/D) | Day 1 to Day 12
  To characterize the Cmax/D of AZD2389 following oral administration of multiple ascending doses in healthy participants, including Japanese participants.
Part B (MAD): Observed lowest concentration before the next dose is administered(Ctrough) | Day 1 to Day 12
  To characterize the Ctrough of AZD2389 following oral administration of multiple ascending doses in healthy participants, including Japanese participants.
Part B (MAD): Individual and cumulative percentage of dose excreted unchanged in urine from time t1 to time t2 [fe(t1-t2)] | Day 1 and Days 10 to 12
  To characterize the fe(t1-t2) of AZD2389 following oral administration of multiple ascending doses in healthy participants, including Japanese participants.
Part B (MAD): Accumulation ratio for AUC (Rac AUC) | Day 1 to Day 12
  To characterize the Rac AUC of AZD2389 following oral administration of multiple ascending doses in healthy participants, including Japanese participants.
Part B (MAD): Accumulation ratio for Cmax (Rac Cmax) | Day 1 to Day 12
  To characterize the Rac Cmax of AZD2389 following oral administration of multiple ascending doses in healthy participants, including Japanese participants.
Part B (MAD): Time to reach peak or maximum observed concentration (tmax) | Day 1 to Day 12
  To characterize the tmax of AZD2389 following oral administration of multiple ascending doses in healthy participants, including Japanese participants.
Part B (MAD): Apparent terminal elimination half-life (t½λz) | Day 1 to Day 12
  To characterize the t½λz of AZD2389 following oral administration of multiple ascending doses in healthy participants, including Japanese participants.
Part B (MAD): Apparent volume of distribution based on the terminal phase (Vz/F) | Day 1 to Day 12
  To characterize the Vz/F of AZD2389 following oral administration of multiple ascending doses in healthy participants, including Japanese participants.
Part B (MAD): Change in PD biomarkers over time | Days 1, 2, 4, 8, and 10
  To characterize the percentage change in PD biomarkers over time compared to baseline of AZD2389 following oral administration of multiple ascending doses in healthy participants, including Japanese participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/